CLINICAL TRIAL: NCT07341295
Title: Percezione Dello Stress e Cultura Della Sicurezza: Analisi Dei Fattori Critici in Ambito Sanitario (SICURES)
Brief Title: Perception of Stress and Safety Culture: Analysis of Critical Factors in Healthcare (SICURES)
Acronym: SICURES
Status: Completed | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Other Study IDs: L2-376
Record Dates: First submitted 2025-12-15; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-07

CONDITIONS: Work Stress; Patient Safety
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthcare professionals: healthcare professionals

SUMMARY:
The study adopts an observational design, based on a sample of 143 healthcare professionals, using two validated anonymous questionnaires: the Perceived Stress Scale (PSS-10) to measure perceived stress levels and the Hospital Survey on Patient Safety Culture 2.0 (SOPS AHRQ) to assess perceptions of patient safety culture.

Data collection will take place at a single point in time and without external intervention, on a sample of healthcare professionals belonging to the various hospital operating units of the CCM.

Objectives (primary and secondary):

* Primary: This study aims to analyze whether the levels of risk management perceived by healthcare professionals are predictive of perceived stress levels in the same clinical context.
* Secondary:

  * Assess the level of stress perceived by healthcare professionals
  * Explore the perception of patient safety culture
  * Analyze the correlation between perceived stress and safety culture in hospital settings
  * Identify possible critical areas or organizational factors that contribute to the onset of stress and influence the perception of safety in care

ELIGIBILITY:
Inclusion Criteria:

* healthcare professionals of CCM DAPS'

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthcare professionals of CCM DAPS'
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
relationship betweemn levels of risk management perceived and perceived stress levels | July 2025 - October 2025
  This study aims to analyze whether the levels of risk management perceived by healthcare professionals are predictive of perceived stress levels in the same clinical context.

CONTACTS AND LOCATIONS:
Locations (1):
- Irrcs Centro Cardiologico Monzino, Milan, MI, Italy